CLINICAL TRIAL: NCT00869557
Title: A Phase 2, Randomized, Double-Blinded Study of the Safety and Efficacy of Elvitegravir/Emtricitabine/Tenofovir Disoproxil Fumarate/GS-9350 Versus Atripla® (Efavirenz 600 mg/Emtricitabine 200 mg/Tenofovir Disoproxil Fumarate 300 mg) in HIV-1 Infected, Antiretroviral Treatment-Naive Adults
Brief Title: Study of the Safety and Efficacy of Stribild Versus Atripla in Human Immunodeficiency Virus, Type 1 (HIV-1) Infected, Antiretroviral Treatment-Naive Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-236-0104
Record Dates: First submitted 2009-03-24; First posted 2009-03-26 (Estimated); Results first posted 2012-10-22 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: HIV; HIV Infections
Keywords: HIV; HIV-1; Antiretroviral Treatment-Naive; treatment naive
MeSH Terms: conditions — HIV Infections | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stribild (Experimental)
  Interventions: Drug: Stribild
- Atripla (Active Comparator)
  Interventions: Drug: Atripla

INTERVENTIONS:
Drug: Stribild — Stribild (EVG 150 mg/COBI 150 mg/FTC 200 mg/TDF 300 mg) STR once daily (QD) + placebo to match Atripla once daily prior to bedtime (QHS)
  Arms: Stribild
Drug: Atripla — Atripla (EFV 150 mg/FTC 200mg/TDF 300 mg) STR QHS + placebo to match Stribild QD
  Arms: Atripla

SUMMARY:
The objective of this double-blinded, multicenter, randomized, active-controlled study is to evaluate the safety and efficacy of Stribild, a single-tablet regimen (STR) containing fixed doses of elvitegravir (EVG)/GS-9350 (cobicistat; COBI)/emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF) versus efavirenz (EFV)/FTC/TDF (Atripla) in HIV-1 infected, antiretroviral treatment-naive adult participants. Stribild offers an alternative STR for patients who are not candidates for non-nucleoside reverse transcriptor (NNRTI)-based STRs.

Participants will be randomized in a 2:1 ratio to receive Stribild or Atripla. Randomization will be stratified by HIV-1 RNA level (≤ 100,000 copies/mL or > 100,000 copies/mL) at screening. After Week 48, participants will continue to take their blinded study drug and attend visits every 12 weeks until treatment assignments are unblinded (Week 60), at which point all participants will attend an Unblinding Visit and be given the option to participate in an open-label rollover extension (the extension is scheduled to be open until Stribild becomes commercially available, or until Gilead Sciences elects to terminate the study).

ELIGIBILITY:
Inclusion Criteria:

* Plasma HIV-1 RNA levels ≥ 5,000 copies/mL
* No prior use of any approved or experimental anti-HIV drug
* Normal electrocardiogram (ECG)
* Adequate renal function: estimated glomerular filtration rate ≥ 80 mL/min according to the Cockcroft-Gault formula
* Hepatic transaminases ≤ 2.5 x upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Adequate hematologic function
* Cluster determinant 4 (CD4) cell count > 50 cells/µL
* Serum amylase ≤ 1.5 x ULN
* Normal thyroid-stimulating hormone
* Negative serum pregnancy test (for females of childbearing potential only)
* Males and females of childbearing potential must agree to utilize highly effective contraception methods from screening throughout the duration of study treatment and for 12 weeks following the last dose of study drugs
* Life expectancy ≥ 1 year
* Ability to understand and sign a written informed consent form

Exclusion Criteria:

* New acquired immunodeficiency syndrome (AIDS)-defining condition diagnosed within the 30 days prior to screening
* Documented drug resistance to nucleoside reverse transcriptase inhibitors or nonnucleoside reverse transcriptase inhibitors or primary protease inhibitor resistance mutation(s)
* Hepatitis B surface antigen positive
* Hepatitis C antibody positive
* Participants experiencing cirrhosis
* Participants experiencing ascites
* Participants experiencing encephalopathy
* Females who are breastfeeding
* Positive serum pregnancy test (for females of childbearing potential)
* Vaccinated within 90 days of study dosing
* History or family history of Long QT Syndrome or family history of sudden cardiac death or unexplained death in an otherwise healthy individual under the age of 30
* Presence or history of cardiovascular disease, cardiomyopathy, and/or cardiac conduction abnormalities
* Prolonged QTcF interval at screening
* PR interval ≥ 200 msec or ≤ 120 msec on ECG at screening
* QRS ≥ 120 msec on ECG at screening
* Implanted defibrillator or pacemaker
* Participants receiving ongoing therapy with any disallowed medications
* Current alcohol or substance use judged to potentially interfere with participant study compliance
* History of or ongoing malignancy (including untreated carcinoma in situ) other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, noninvasive cutaneous squamous carcinoma
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline
* Participation in any other clinical trial without prior approval
* Medications contraindicated for use with EFV, EVG, COBI, FTC, or TDF
* Any known allergies to the excipients of Atripla or Stribild tablets
* Any other clinical condition or prior therapy that would make the participant unsuitable for the study or unable to comply with the dosing requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Health for Life Clinic, PLLC, Little Rock, Arkansas
  - The Living Hope Foundation, Long Beach, California
  - Peter J. Ruane, MD, Inc., Los Angeles, California
  - Orange Coast Medical Group, Newport Beach, California
  - East Bay AIDS Center, Oakland, California
  - Metropolis Medical, San Francisco, California
  - Apex Research Institute, Denver, Colorado
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - Capital Medical Associates PC, Washington D.C., District of Columbia
  - Broward Health, Fort Lauderdale, Florida
  - Gary Richmond, MD, PA, Inc., Fort Lauderdale, Florida
  - Wohlfeiler, Piperato and Associates, LLC, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Infectious Disease of Central Florida, Orlando, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - Infectious Disease Specialists of Atlanta (IDSA), Decatur, Georgia
  - Northstar Medical Center, Chicago, Illinois
  - Chase Brexton Health Services, Inc., Baltimore, Maryland
  - Community Research Initiative of New England, Boston, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Southampton Healthcare, Inc., St Louis, Missouri
  - Southwest C.A.R.E. Center, Santa Fe, New Mexico
  - Chelsea Village Medical, New York, New York
  - Ricky K. Hsu, MD, PC, New York, New York
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - Nicholaos Bellos, MD, PA, Dallas, Texas
  - AIDS Arms/ Peabody Health Center, Dallas, Texas
  - Gordon E. Crofoot, MD, PA, Houston, Texas
  - TribalMed, Seattle, Washington

REFERENCES:
- [Result] Cohen C, Elion R, Ruane P, Shamblaw D, DeJesus E, Rashbaum B, Chuck SL, Yale K, Liu HC, Warren DR, Ramanathan S, Kearney BP. Randomized, phase 2 evaluation of two single-tablet regimens elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate versus efavirenz/emtricitabine/tenofovir disoproxil fumarate for the initial treatment of HIV infection. AIDS. 2011 Mar 27;25(6):F7-12. doi: 10.1097/QAD.0b013e328345766f. PMID 21412057
- See also: Gilead Sciences — http://www.gilead.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in a total of 30 sites in the United States. The first participant was screened on 30 March 2009.
  Last participant visit:
  * Primary endpoint analysis (Week 24): November 2009
  * Week 48 analysis: April 2010
  * Week 96 analysis: March 2011
  * End of study: September 2013
Pre-assignment Details: 126 participants were screened; 71 were randomized (48 to the Stribild group and 23 to the Atripla group). All randomized participants received at least 1 dose of study medication and comprised the safety and intent-to-treat (ITT) analysis sets. No site enrolled more than 7% of participants.
Groups:
- Stribild: Stribild (elvitegravir [EVG] 150 mg/GS-9350 [cobicistat; COBI] 150 mg/emtricitabine [FTC] 200 mg/tenofovir disoproxil fumarate [TDF] 300 mg) once daily (QD) and placebo to match Atripla once daily prior to bedtime (QHS) were administered during the double-blind phase. Stribild QD was administered during the extension phase.
- Atripla: Atripla (efavirenz [EFV] 150 mg/FTC 200 mg/TDF 300 mg) QHS and placebo to match Stribild QD were administered during the double blind phase. Stribild QD was administered during the extension phase.
Period: Randomized Phase
Arm/Group | Stribild | Atripla
Started | 48 | 23
Completed | 45 | 21
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Investigator's Discretion | 1 | 0
Not completed — Withdrew Consent | 0 | 1
Period: Extension Phase
Arm/Group | Stribild | Atripla
Started | 45 | 14 (Seven participants completing randomized Atripla treatment did not enter open-label extension phase.)
Completed | 35 | 11
Not Completed | 10 | 3
Not completed — Adverse Event | 2 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Investigator's Discretion | 2 | 0
Not completed — Withdrew Consent | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants were randomized and received at least 1 dose of study medication.
Groups:
- Stribild: Stribild QD and placebo to match Atripla QHS were administered during the double-blind phase. Stribild QD was administered during the extension phase.
- Atripla: Atripla QHS and placebo to match Stribild QD were administered during the double blind phase. Stribild QD was administered during the extension phase.
- Total: Total of all reporting groups
Arm/Group | Stribild | Atripla | Total
Number analyzed (Participants) | 48 | 23 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 23 | 71
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (8.9) | 35 (9.6) | 36 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 44 | 21 | 65
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Black | 12 | 5 | 17
  White | 33 | 18 | 51
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 48 | 23 | 71
HIV Disease Status [Number; unit: participants]
  Asymptomatic | 40 | 22 | 62
  Symptomatic HIV Infections | 5 | 0 | 5
  AIDS | 3 | 1 | 4
Hepatitis B Virus (HBV) Infection Status [Number; unit: participants]
  Negative | 48 | 23 | 71
  Positive | 0 | 0 | 0
Hepatitis C Virus (HCV) Infection Status [Number; unit: participants]
  Negative | 48 | 23 | 71
  Positive | 0 | 0 | 0
HIV-1 RNA Category (copies/mL) [Number; unit: participants]
  ≤ 100,000 | 37 | 18 | 55
  > 100,000 | 11 | 5 | 16
Cluster Determinant 4 (CD4) Cell Count (/µL) [Number; unit: participants]
  ≤ 50 | 0 | 0 | 0
  51 to ≤ 200 | 7 | 0 | 7
  201 to ≤ 350 | 17 | 8 | 25
  351 to ≤ 500 | 14 | 5 | 19
  > 500 | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With HIV-1 Ribonucleic Acid (RNA) Less Than 50 Copies/mL at Week 24
Description: The percentage of participants with plasma HIV-1 RNA < 50 copies/mL at Week 24 was summarized.
Time Frame: Week 24
Population: ITT analysis set (all participants who were randomized into the study and received at least 1 dose of study drug). The missing = failure (M = F) analysis method was used in which all missing data were considered as failure (HIV-1 RNA ≥ 50 copies/mL).
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | Atripla
Number analyzed (Participants) | 48 | 23
percentage of participants | 89.6 | 87.0
Statistical Analysis 1: Comparison: Stribild vs Atripla; The null hypothesis was that the response rate (proportion of participants with HIV-1 RNA < 50 copies/mL at Week 24) in the Stribild group was at least 12% worse than the response rate in Atripla group; the alternative hypothesis was that the response rate in the Stribild group was less than 12% worse than that in the Atripla group; Test type: Non-Inferiority or Equivalence — A total sample size of 75 participants randomized in a 2:1 ratio had 26% power to evaluate noninferiority with respect to the response rate of HIV-1 RNA < 50 copies/mL at Week 24 if a response rate of 84% for both treatment groups and a noninferiority margin of 0.12 were assumed. A total of 71 participants were enrolled in the study (4 fewer than planned); Difference in the response rates (%) = 2.8, 95% CI 2-sided [-14.5 to 20.1] — The 95% confidence interval was computed using normal approximation stratified by baseline HIV-1 RNA stratum (≤ 100,000 or > 100,000 copies/mL)

2. Secondary Outcome: The Percentage of Participants With HIV-1 RNA Less Than 50 Copies/mL at Week 48
Description: The percentage of participants with plasma HIV-1 RNA < 50 copies/mL at Week 48 was summarized.
Time Frame: Week 48
Population: ITT analysis set; M = F analysis (all missing data were considered as failure [HIV-1 RNA ≥ 50 copies/mL]).
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | Atripla
Number analyzed (Participants) | 48 | 23
percentage of participants | 89.6 | 87.0

3. Secondary Outcome: Change From Baseline in HIV-1 RNA (log_10 Copies/mL)
Description: Change = Week 24 or 48 value minus baseline value
Time Frame: Baseline to Weeks 24 and 48
Population: ITT analysis set; The missing = excluded (M = E) analysis method was used in which all missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: log_10 copies/mL
Arm/Group | Stribild | Atripla
Number analyzed (Participants) | 45 | 21
log_10 copies/mL
  Baseline to Week 24 | -2.87 (0.578) | -2.88 (0.586)
  Baseline to Week 48 | -2.89 (0.570) | -2.71 (0.933)

4. Secondary Outcome: Change From Baseline in Cluster Determinant 4 (CD4) Cell Count at Week 24
Description: Change = Week 24 value minus baseline value
Time Frame: Baseline to Week 24
Population: ITT analysis set. M = E analysis (all missing data were excluded from the analysis).
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Stribild | Atripla
Number analyzed (Participants) | 44 | 21
cells/µL | 161 (141.1) | 117 (143.7)

5. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 48
Description: Change = Week 48 value minus baseline value
Time Frame: Baseline to Week 48
Population: ITT analysis set; M = E analysis (all missing data were excluded from the analysis).
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Stribild | Atripla
Number analyzed (Participants) | 45 | 21
cells/µL | 240 (172.8) | 166 (158.5)

6. Secondary Outcome: The Percentage of Participants With Virologic Success at Weeks 24 and 48 Using FDA-Defined Snapshot Analysis and HIV-1 RNA Less Than 50 Copies/mL
Description: The percentage of participants with virologic success at Weeks 24 and 48 assessed using the FDA-defined snapshot analysis for an HIV-1 RNA cutoff of 50 copies/mL was summarized.
Time Frame: Baseline to Weeks 24 and 48
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | Atripla
Number analyzed (Participants) | 48 | 23
percentage of participants
  Virologic Success at Week 24 | 89.6 | 87.0
  Virologic Success at Week 48 | 91.7 | 82.6

ADVERSE EVENTS:
Time Frame: Adverse events are reported for the double-blind treatment period (up to 60 weeks) for the randomized treatment group (Stribild and Atripla), and for the double-blind and open-label period (up to 224 weeks) for the All Stribild group.
Groups:
- Stribild: Stribild and placebo to match Atripla were administered during the double-blind phase.
- Atripla: Atripla QHS and placebo to match Stribild QD were administered during the double blind phase.
- All Stribild: The All Stribild safety analysis set included all participants who received at least 1 dose of Stribild in the randomized phase or in the open-label extension phase. Adverse event data presented in this group include the following: Adverse events collected from participants who were initially randomized to the double-blind Stribild group while they received double-blind Stribild during the randomized phase and open-label Stribild during the extension phase; adverse events collected from the open-label Stribild extension phase only from the participants who were initially randomized to the Atripla group during the randomized phase.
Arm/Group | Stribild | Atripla | All Stribild
Serious Adverse Events (participants affected / at risk) | 2/48 | 1/23 | 9/62
Other Adverse Events (participants affected / at risk) | 39/48 | 20/23 | 57/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stribild (N=48) | Atripla (N=23) | All Stribild (N=62)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 2
Staphylococcal infection (Infections and infestations) | 1 | 0 | 1
Vaccination site cellulitis (Infections and infestations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 3
Hepatitis C (Infections and infestations) | 0 | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 1
Acute hepatitis C (Infections and infestations) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stribild (N=48) | Atripla (N=23) | All Stribild (N=62)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1
Conjunctivitis (Eye disorders) | 1 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 13 | 4 | 16
Nausea (Gastrointestinal disorders) | 4 | 2 | 5
Abdominal distension (Gastrointestinal disorders) | 3 | 1 | 5
Flatulence (Gastrointestinal disorders) | 3 | 1 | 4
Vomiting (Gastrointestinal disorders) | 2 | 2 | 3
Fatigue (General disorders) | 8 | 4 | 11
Pain (General disorders) | 3 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 4 | 6 | 17
Bronchitis (Infections and infestations) | 6 | 2 | 15
Nasopharyngitis (Infections and infestations) | 2 | 2 | 5
Urinary tract infection (Infections and infestations) | 3 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 7
Headache (Nervous system disorders) | 7 | 4 | 11
Somnolence (Nervous system disorders) | 2 | 2 | 2
Dizziness (Nervous system disorders) | 0 | 3 | 1
Abnormal dreams (Psychiatric disorders) | 5 | 8 | 5
Insomnia (Psychiatric disorders) | 6 | 2 | 10
Depression (Psychiatric disorders) | 4 | 2 | 11
Anxiety (Psychiatric disorders) | 2 | 3 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 12
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 5 | 4 | 8
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 0 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 4
Sinusitis (Infections and infestations) | 2 | 5 | 12
Syphilis (Infections and infestations) | 3 | 0 | 9
Folliculitis (Infections and infestations) | 2 | 0 | 5
Influenza (Infections and infestations) | 2 | 0 | 5
Oral herpes (Infections and infestations) | 2 | 1 | 5
Pharyngitis (Infections and infestations) | 1 | 0 | 5
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 5
Urethritis (Infections and infestations) | 1 | 1 | 6
Onychomycosis (Infections and infestations) | 1 | 0 | 5
Papilloma viral infection (Infections and infestations) | 2 | 0 | 4
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 6
Anorectal human papilloma virus infection (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 5
Paraesthesia (Nervous system disorders) | 1 | 0 | 4
Proteinuria (Renal and urinary disorders) | 2 | 0 | 4
Epididymitis (Reproductive system and breast disorders) | 0 | 0 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 4
Hypertension (Vascular disorders) | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years